CLINICAL TRIAL: NCT05681793
Title: Survey on the Clinical Assessment of the Psychological Status of a Patient Over 75 Years Old in Oncology During the Realization of the G8 Score
Brief Title: Survey on the Clinical Assessment of the Psychological Status of a Patient Over 75 Years Old in Oncology During the Realization of the G8 Score (CADEPO)
Acronym: CADEPO
Status: Completed | Type: Observational
Sponsor: Hopital Nord Franche-Comte (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A02329-34
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to make a statement concerning the identification of depressive symptoms at the time of the realization of the G8 score in patients over 75 with cancer and followed in oncology.

The main question it aims to answer are:

* Compare the medical hetero-evaluation of depressive symptoms via the G8 "neuro-psychiatric disorders" item score with a self-evaluation via the GDS-15 score
* Evaluate the number of patients over 75 treated with antidepressants
* Evaluate the proportion of patients with depressive symptoms according to the predisposing factors
* Compare the number of patients followed in oncogeriatrics over the period from 01/01/2022 to 02/28/2022 and the period from 01/01/2023 to 02/28/2023

Participants will complete a self-questionnaire (GDS-15 score) as well as a socio-demographic sheet.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 75 and over
* Patients receiving treatment at the day hospital or oncology week hospital
* Patients informed and having not presented any opposition to their participation

Exclusion Criteria:

* Patients under the age of 75
* Patients under guardianship or curatorship
* Patients without social security
* Cognitive disorders compromising the understanding of the information and the performance of the study (in particular the completion of a self-administered questionnaire), in the opinion of the oncologist

Ages: 75 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients over 75 presenting eligibility criteria and undergoing oncological treatment and coming for consultation in the Hôpital Nord Franche-Comté
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-03-02 (Actual); Study Completion 2023-04-02 (Actual)

PRIMARY OUTCOMES:
Comparison the medical hetero-evaluation of depressive symptoms via the G8 "neuro-psychiatric disorders" item score with a self-evaluation via the GDS-15 score, in patients over 75 years of age with cancer and follow-up in oncology | 2 months
  Difference between the evaluation of the health professionals of the item "Neuropsychiatric problems" of the G8 score (no depression versus moderate or severe depression) and the responses of the patients to the self-administered questionnaire GDS-15 (Geriatric Depression Scale) ( 0 to 4: normal versus 5 to 15: moderate to severe depression).

SECONDARY OUTCOMES:
Evaluation of the number of patients over 75 on antidepressants included in this study | 2 months
  Percentage of patients included in this study and being treated with antidepressants
Evaluation of the proportion of patients with depressive symptoms according to the predisposing factors with a sociodemographic sheet and from the medical file | 2 months
  Percentage of patients with depressive symptoms according to the predisposing factors (age, gender, housing in urban or rural areas,distance (in travel time) between the oncology department and home, social isolation, income, marital status, socio-professional category, type of cancer), taken from a sociodemographic sheet distributed to the patient and from the medical file
Compare the number of patients followed in oncogeriatrics over the period from 01/01/22 to 02/28/22 and the period from 01/01/2023 to 02/28/2023 | 2 months
  Percentage of patients followed in oncogeriatrics over the period from 01/01/2022 to 02/28/2022 and the period from 01/01/2023 to 02/28/2023

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Nord Franche-Comté, Trévenans, France

IPD SHARING:
Plan to Share IPD: No